CLINICAL TRIAL: NCT02303704
Title: Myocardial Protection With Multiport Antegrade Cold Blood Cardioplegia and Continuous Controlled Warm Shot Through Vein Grafts During Proximal Ends Anastomosis in Conventional CABG
Brief Title: Myocardial Protection With Multiport Antegrade Cold Blood Cardioplegia
Acronym: MACBC
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Chaudhry Pervaiz Elahi Institute of Cardiology (Other Government)
Responsible Party: Principal Investigator, Muhammad Sher-i-Murtaza, senior registrar cardiac surgery, Multan institute of cardiology, multan, pakistan., Chaudhry Pervaiz Elahi Institute of Cardiology
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: multanic
Record Dates: First submitted 2014-11-19; First posted 2014-12-01 (Estimated); Results first posted 2014-12-08 (Estimated); Last update posted 2021-02-09 (Actual); Status verified 2021-02

CONDITIONS: Coronary Artery Bypass Surgery
Keywords: Multiperfusion set; Myocardial protection; Coronary Artery Bypass Grafting

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- multiport antegrade cardioplegia (Active Comparator): Patients who received multiport antegrade cardioplegia and continuous controlled warm blood perfusion through vein grafts.
  Interventions: Procedure: multiport antegrade cardioplegia
- Aortic root antegrade cardioplegia (Active Comparator): Patients who underwent routine conventional CABG with antegrade aortic root cardioplegia without warm blood perfusion
  Interventions: Procedure: Aortic root antegrade cardioplegia

INTERVENTIONS:
Procedure: multiport antegrade cardioplegia — Cold blood cardioplegia was used for myocardial protection and just before the removal of the aortic cross-clamp, warm blood shot (normo-kalemic) was started through multi-perfusion set attached to cardioplegia cannula in the aortic root and vein grafts.As contraction of heart started the multiport limb attached to cardioplegia cannula was off and cross clamp was removed .The warm perfusion through the vein grafts was continued at controlled pressures of about 50-70 mmHg, flow rate of 10-30ml/min/graft and temperature of 35-37 oC
  Other Names: multiperfusion set
  Arms: multiport antegrade cardioplegia
Procedure: Aortic root antegrade cardioplegia — only cold blood cardioplegia was used for myocardial protection without hotshot.
  Arms: Aortic root antegrade cardioplegia

SUMMARY:
In spite improvements in methods of myocardial protection, peri-operative myocardial damage is still the commonest cause of early morbidity and mortality after technically successful CABG Surgery. What is the optimum method of myocardial protection is still debatable.

The investigators conducted this study to see effects of multiport antegrade cold blood cardioplegia on myocardial protection, along with continuous controlled warm blood perfusion through veins graft during proximal ends anastomosis in conventional CABG surgery in patients having multi-vessel disease.

DETAILED DESCRIPTION:
A prospective randomized controlled study was conducted between April-2013 and June-2014, in the Department of Cardiac Surgery, Chaudary Pervaiz Elahi Institute of cardiology (CPEIC) Multan, Pakistan. The CPEIC is a tertiary cardiac care center and is presently performing over 600 coronary artery bypass surgery annually. The study was conducted in strict compliance of the rules established by the revised Helsinki convention and had approval from the ethical committee of the institute.

Patients undergoing isolated conventional CABG were included in the study except; The redo CABG, those who required 2 or less than 2 grafts, patients who had major postoperative neurological complications like stroke, 2nd arterial graft along with LIMA, patients who need CABG within a week of STEMI or NSTEMI and Patients with calcified or diseased aorta in which single cross clamp technique was used for proximal aorto-coronary anastomosis.

The patients were randomized into two groups by using draw randomization technique. The investigators made 112 sets, each set containing four patients. The staff nurse on duty was requested to pick up the two folded papers from four containing hidden identity of the patients. The patients chosen by draw were included in the study group, others in the control group.

Group I: Patients who received multiport antegrade cardioplegia and continuous controlled warm blood perfusion through vein grafts (Study Group) and Group II: Patients who underwent routine conventional CABG with antegrade aortic root cardioplegia without warm blood perfusion (Control Group).

All operations were carried out by two consultant surgeons at the investigators institution, who are certified cardiac surgeons with sufficient experience. Patients were premedicated with oral dose of 3mg bromazepam the night before surgery. Anaesthesia was induced with intra-venous morphine (0.1mg/kg), midazolam (0.05-0.1 mg /kg), and propofol (1.0-2.5 mg/kg titrated according to the response. They were given atracuronium (1mg/kg) before endotracheal intubation. The anaesthesia was maintained with sevoflorane/isoflurane.

In all patients the standard cardiopulmonary bypass (CPB) was established with an ascending aortic arterial cannula and a two stage single venous cannula in the right atrium. The CPB circuit was primed with crystalloid Ringer's solution. Heparin was administered in a dose of 400 U/Kg. The body temperature was lowered to 30-32°C. The local cooling was achieved with ice cold saline. Cold blood cardioplegia was used in each group. The first dose of cardioplegia was 10-15 ml/kg and further doses were given as 5-7ml/kg repeated after each graft or after 20 minutes. Cold blood cardioplegia was given by using cardioplegia delivery system including heat exchanger in both groups. A cardioplegia delivery cannula with a separate vent line (DLP Medtronic, Grand Rapids, MI, USA) was inserted into the ascending aorta. The pump flow rate was kept between 2.0 and 2.4 L/min/m2 to maintain a mean arterial pressure of 55 - 70 mmHg. In both groups, myocardial protection was achieved by an initial antegrade infusion of cold (4 °C) blood cardioplegic potassium solution followed by intermittent antegrade cold blood cardioplegia at the completion of each distal anastomosis via a cardioplegia delivery cannula from the aortic root. Whereas in Group I, a multiple perfusion set was used to deliver cardioplegia simultaneously in aortic root and vein grafts. After the distal anastomosis of each vein graft had been completed, the proximal ends were connected to the free branch of the multi- perfusion set. In this way, simultaneous intermittent antegrade graft cardioplegia was administered in addition to aortic root cardioplegia (named as multiport antegrade cardioplegia).

LIMA and great saphenous vein were used as conduits. LIMA was anastomosed to LAD and other coronary vessels received greater saphenous vein grafts as conduits.

Just before the removal of the aortic cross-clamp, warm blood shot (normo-kalemic) was started through multi-perfusion set attached to cardioplegia cannula in the aortic root and vein grafts in Group I. As contraction of heart started the multiport limb attached to cardioplegia cannula was off and cross clamp was removed .The warm perfusion through the vein grafts was continued at controlled pressures of about 50-70 mmHg, flow rate of 10-30ml/min/graft and temperature of 35-37 oC. Proximal anastmosis was performed in both groups using partial occluding clamp.

The necessity of inotropic support and the choice of inotropic drugs to be administered during weaning from cardiopulmonary bypass (CPB) were determined by a cardiac anaesthetist team, who were blinded and independent with respect to the study.

The CK-MB levels were determined at five points of time i.e. before operation, immediately after shifting to ICU, at 12, 24 hours and 36 hours after shifting of patient to ICU. The reagent used for determining the serum CK-MB levels was the product of Merck (Merck, France) and the designated reference value for detection of myocardial damage were >25 units/liter for CK-MB.

448 patient characteristics were prospectively entered in the investigators electronic database (CASCADE DATABASES, Lahore, Pakistan). The study specific data not included in the database were separately entered in a Microsoft Excel spreadsheet (MS Excel, version 2007, Microsoft Co USA). The statistical analysis was carried out using SPSS (SPSS version 20, SPSS Inc, Chicago, IL). The preoperative, operative and postoperative characteristics were summarized using means and standard deviation for the numeric variables. The groups were compared using Student's t-test for numeric variables and Chi-square test for categorical variables.

The significance of differences between the groups was expressed as p-value and a value of <0.05 was considered significant.

ELIGIBILITY:
Inclusion Criteria:

* All patients undergoing isolated conventional CABG were included in the study

Exclusion Criteria:

The redo CABG surgery. Those who required 2 or less than 2 grafts. Patients who had major postoperative neurological complications like stroke. 2nd arterial graft along with LIMA. Patients who need CABG within a week of STEMI or NSTEMI. Patients with calcified or diseased aorta in which single cross clamp technique was used for proximal aorto-coronary anastomosis

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 448 (Actual)
Dates: Start 2013-04; Primary Completion 2014-06 (Actual); Study Completion 2014-08 (Actual)

REFERENCES:
- [Background] Mack MJ, Brown PP, Kugelmass AD, Battaglia SL, Tarkington LG, Simon AW, Culler SD, Becker ER. Current status and outcomes of coronary revascularization 1999 to 2002: 148,396 surgical and percutaneous procedures. Ann Thorac Surg. 2004 Mar;77(3):761-6; discussion 766-8. doi: 10.1016/j.athoracsur.2003.06.019. PMID 14992867
- [Background] Onorati F, De Feo M, Mastroroberto P, Cristodoro L, Pezzo F, Renzulli A, Cotrufo M. Determinants and prognosis of myocardial damage after coronary artery bypass grafting. Ann Thorac Surg. 2005 Mar;79(3):837-45. doi: 10.1016/j.athoracsur.2004.07.060. PMID 15734390
- [Background] Steuer J, Horte LG, Lindahl B, Stahle E. Impact of perioperative myocardial injury on early and long-term outcome after coronary artery bypass grafting. Eur Heart J. 2002 Aug;23(15):1219-27. doi: 10.1053/euhj.2002.3171. PMID 12127924
- [Background] Soltesz EG, Laurence RG, De Grand AM, Cohn LH, Mihaljevic T, Frangioni JV. Image-guided quantification of cardioplegia delivery during cardiac surgery. Heart Surg Forum. 2007;10(5):E381-6. doi: 10.1532/HSF98.20071099. PMID 17855203
- [Background] Sanjay OP, Srikrishna SV, Prashanth P, Kajrekar P, Vincent V. Antegrade versus antegrade with retrograde delivery of cardioplegic solution in myocardial revascularisation. A clinical study in patients with triple vessel coronary artery disease. Ann Card Anaesth. 2003 Jul;6(2):143-8. PMID 17827576
- [Background] Teoh KH, Christakis GT, Weisel RD, Fremes SE, Mickle DA, Romaschin AD, Harding RS, Ivanov J, Madonik MM, Ross IM, et al. Accelerated myocardial metabolic recovery with terminal warm blood cardioplegia. J Thorac Cardiovasc Surg. 1986 Jun;91(6):888-95. PMID 3520161
- [Background] Onorati F, Renzulli A, De Feo M, Santarpino G, Gregorio R, Biondi A, Cerasuolo F, Cotrufo M. Does antegrade blood cardioplegia alone provide adequate myocardial protection in patients with left main stem disease? J Thorac Cardiovasc Surg. 2003 Nov;126(5):1345-51. doi: 10.1016/s0022-5223(03)00736-0. PMID 14666005
- [Background] Tian G, Xiang B, Dai G, Sun J, Lindsay WG, Deslauriers R. Simultaneous antegrade/retrograde cardioplegia protects myocardium distal to a coronary occlusion: a study in isolated pig hearts. Magn Reson Med. 2001 Oct;46(4):773-80. doi: 10.1002/mrm.1256. PMID 11590654
- [Background] Allen BS, Winkelmann JW, Hanafy H, Hartz RS, Bolling KS, Ham J, Feinstein S. Retrograde cardioplegia does not adequately perfuse the right ventricle. J Thorac Cardiovasc Surg. 1995 Jun;109(6):1116-24; discussion 1124-6. doi: 10.1016/S0022-5223(95)70195-8. PMID 7776676
- [Background] Ardehali A, Gates RN, Laks H, Drinkwater DC Jr, Rudis E, Sorensen TJ, Chang P, Aharon A. The regional capillary distribution of retrograde blood cardioplegia in explanted human hearts. J Thorac Cardiovasc Surg. 1995 May;109(5):935-9; discussion 939-40. doi: 10.1016/S0022-5223(95)70319-5. PMID 7739255
- [Background] Carrier M, Gregoire J, Khalil A, Thai P, Latour JG, Pelletier LC. Myocardial distribution of retrograde cardioplegic solution assessed by myocardial thallium 201 uptake. J Thorac Cardiovasc Surg. 1994 Dec;108(6):1115-8. PMID 7983880
- [Background] Sabzi F, Zokaei A. Factors predicting coronary sinus rupture following cannula insertion for retrograde cardioplegia. Clin Med Insights Cardiol. 2012;6:1-6. doi: 10.4137/CMC.S7861. Epub 2011 Dec 6. PMID 22259260
- [Background] Panos AL, Ali IS, Birnbaum PL, Barrozo CA, al-Nowaiser O, Salerno TA. Coronary sinus injuries during retrograde continuous normothermic blood cardioplegia. Ann Thorac Surg. 1992 Dec;54(6):1137-8. doi: 10.1016/0003-4975(92)90082-f. PMID 1449299
- [Background] Radmehr H, Soleimani A, Tatari H, Salehi M. Does combined antegrade-retrograde cardioplegia have any superiority over antegrade cardioplegia? Heart Lung Circ. 2008 Dec;17(6):475-7. doi: 10.1016/j.hlc.2008.04.009. Epub 2008 Jul 26. PMID 18676202
- [Result] Guyton RA, Thourani VH, Puskas JD, Shanewise JS, Steele MA, Palmer-Steele CL, Vinten-Johansen J. Perfusion-assisted direct coronary artery bypass: selective graft perfusion in off-pump cases. Ann Thorac Surg. 2000 Jan;69(1):171-5. doi: 10.1016/s0003-4975(99)01386-7. PMID 10654508
- [Result] Lu F, Ji BY, Liu JP, Liu MZ, Wang GY, Hu SS. Passive graft perfusion in off-pump coronary artery bypass grafting. Chin Med J (Engl). 2007 Feb 5;120(3):192-6. PMID 17355820
- [Result] Vassiliades TA Jr, Nielsen JL, Lonquist JL. Coronary perfusion methods during off-pump coronary artery bypass: results of a randomized clinical trial. Ann Thorac Surg. 2002 Oct;74(4):S1383-9. doi: 10.1016/s0003-4975(02)03912-7. PMID 12400822
- [Result] Goldman BS, Ovil Y, Mycyk T. A technique for selective graft perfusion during aortocoronary bypass. J Card Surg. 1987 Dec;2(4):495-8. doi: 10.1111/j.1540-8191.1987.tb00206.x. PMID 2979995
- [Result] Onem G, Sacar M, Baltalarli A, Ozcan AV, Gurses E, Sungurtekin H. Comparison of simultaneous antegrade/vein graft cardioplegia with antegrade cardioplegia for myocardial protection. Adv Ther. 2006 Nov-Dec;23(6):869-77. doi: 10.1007/BF02850208. PMID 17276955
- [Result] Gürsoy M, Bakuy V, Hatemi AC. Delivering Cardioplegia Beyond Totally Occluded Native Coronary Arteries Through the Saphenous Bypass Vein Graft: Is It Really a Protective Technique? Kosuyolu Kalp Derg. 2012;15:100 -104
- [Result] Hatemi AC, Ulusoy RfE, Gürsoy M, Tongut A. Myocardial Protection with Simultaneous Antegrade/Vein Graft Cardioplegia Compared to Antegrade Cardioplegia Alone in Elective Coronary Artery Bypass Grafting Patients. Balkan Medical Journal. 2011
- [Result] Goncu MT, Sezen M, Toktas F, Ari H, Gunes M, Tiryakioglu O, Yavuz S. Effect of antegrade graft cardioplegia combined with passive graft perfusion in on-pump coronary artery bypass grafting. J Int Med Res. 2010 Jul-Aug;38(4):1333-42. doi: 10.1177/147323001003800415. PMID 20926006

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Multiport Antegrade Cardioplegia | Aortic Root Antegrade Cardioplegia
Started | 220 | 228
Completed | 215 | 219
Not Completed | 5 | 9
Not completed — Protocol Violation | 5 | 9

BASELINE CHARACTERISTICS:
Population: All patients who was enrolled for trial age and gender was clearly defined and noted
Groups:
- Total: Total of all reporting groups
Arm/Group | Multiport Antegrade Cardioplegia | Aortic Root Antegrade Cardioplegia | Total
Number analyzed (Participants) | 215 | 219 | 434
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.97 (8.44) | 53.62 (9.60) | 54.29 (9.06)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 29 | 27 | 56
  Male | 186 | 192 | 378

OUTCOME MEASURES:

1. Primary Outcome: Post-op CK-MB Levels
Description: CK-MB is a marker of Myocardial Damage.
Time Frame: 36 hours after surgery.
Population: All patients in whom Peak CKMB levels were noted within 24 hours after surgery
Measure: Mean (Standard Deviation); unit: IU/L
Arm/Group | Multiport Antegrade Cardioplegia | Aortic Root Antegrade Cardioplegia
Number analyzed (Participants) | 215 | 219
IU/L | 71.70 (41.50) | 92.66 (88.10)
Statistical Analysis 1: Comparison: Multiport Antegrade Cardioplegia vs Aortic Root Antegrade Cardioplegia; Null hypothesis was there is no significant difference between the means of two groups; Test type: Non-Inferiority or Equivalence — to check the equality of means; p < 0.05, t-test, 2 sided — P-value less than 0.05 was considered significant; two compare two independent quantitative groups

2. Secondary Outcome: Pharmacologic Inotropic Support (Adrenaline)
Description: The need, dose and duration of adrenaline infusion to maintain hemodynamic stability after surgery were noted.
Time Frame: Upto 1 week after sugery
Population: All patients in whom Adrenaline was used to wean off the patients from Cardiopulmonary Bypass.
Measure: Mean (Standard Deviation); unit: ug/kg/min
Arm/Group | Multiport Antegrade Cardioplegia | Aortic Root Antegrade Cardioplegia
Number analyzed (Participants) | 215 | 219
ug/kg/min | 0.047 (0.018) | 0.064 (0.82)
Statistical Analysis 1: Comparison: Multiport Antegrade Cardioplegia vs Aortic Root Antegrade Cardioplegia; Test type: Non-Inferiority or Equivalence — to check the equality of means between the two groups; p < 0.05, t-test, 2 sided

3. Secondary Outcome: Pharmacological Inotropic Support (Nor-adrenaline)
Description: The need, dose and duration of Nor-adrenaline infusion to maintain hemodynamic stability after surgery.
Time Frame: Upto 1 week after sugery
Population: All patients in whom Nor-adrenaline was used to wean off the patients from Cardiopulmonary Bypass.
Measure: Mean (Standard Deviation); unit: ug/kg/min
Arm/Group | Multiport Antegrade Cardioplegia | Aortic Root Antegrade Cardioplegia
Number analyzed (Participants) | 215 | 219
ug/kg/min | 0.035 (0.016) | 0.089 (0.50)
Statistical Analysis 1: Comparison: Multiport Antegrade Cardioplegia vs Aortic Root Antegrade Cardioplegia; Null Hypothesis: The dose of nor-adrenaline on weaning from CPB is same for Group I and II; Test type: Non-Inferiority or Equivalence — to check the equality of means; p < 0.05, t-test, 2 sided — p-value <0.05 was considered significant; To compare the means between the two groups, to find out the significant difference between Group I and II

4. Secondary Outcome: Pharamacological Inotropic Support (Dobutamine)
Description: The Need, Dose and duration of Dobutamine to maintain hemodynamic stability after surgery.
Time Frame: Upto 1 week after sugery
Population: All patients in whom Dobutamine was used to wean off the patients from Cardiopulmonary Bypass.
Measure: Mean (Standard Deviation); unit: ug/kg/min
Arm/Group | Multiport Antegrade Cardioplegia | Aortic Root Antegrade Cardioplegia
Number analyzed (Participants) | 215 | 219
ug/kg/min | 3.41 (1.70) | 4.20 (2.24)
Statistical Analysis 1: Comparison: Multiport Antegrade Cardioplegia vs Aortic Root Antegrade Cardioplegia; Test type: Non-Inferiority or Equivalence — to chek the equality of means between the two groups; p < 0.05, t-test, 2 sided

5. Secondary Outcome: Intra-aortic Balloon Pump Counter-pulsation (IABPC) Support
Description: The need of IABPC (mechanical support) before surgery or during weaning from Cardiopulmonary bypass and in ICU to assist in maintaining hemodynamics of the patient.
Time Frame: 24 hours before surgery and upto 1 week of surgical procedure.
Population: All patients who underwent surgery and for whom IABP support was required.
Measure: Number; unit: participants
Arm/Group | Multiport Antegrade Cardioplegia | Aortic Root Antegrade Cardioplegia
Number analyzed (Participants) | 215 | 219
participants | 4 | 14
Statistical Analysis 1: Comparison: Multiport Antegrade Cardioplegia vs Aortic Root Antegrade Cardioplegia; Null Hypothesis:The proportion of IABP use is same between the two groups; Test type: Superiority or Other; p < 0.05, Chi-squared — p- value less than 0.05 was considered as significant difference in proportion between the two groups; two compare the qualitative data between two groups

6. Secondary Outcome: Operative Mortality
Description: Deaths due to surgical complication during or after surgery.
Time Frame: Within 30 days after surgical Procedure
Population: all patients who underwent surgery and monitored for death due to surgical complication.
Measure: Number; unit: participants
Arm/Group | Multiport Antegrade Cardioplegia | Aortic Root Antegrade Cardioplegia
Number analyzed (Participants) | 215 | 219
participants | 1 | 9
Statistical Analysis 1: Comparison: Multiport Antegrade Cardioplegia vs Aortic Root Antegrade Cardioplegia; Null Hypothesis: Operative mortality ratio is same in both groups; Test type: Superiority or Other; p < 0.05, Fisher Exact — P-value <0.05 was considered to be significant i.e. operative mortality is not same between the two groups; Fisher exact test was used because 1 cell (25%) have expected count less than 5

ADVERSE EVENTS:
Time Frame: 1 month after surgery
Description: Adverse event was considered as any complication that will be the direct result of technique used for myocardial protection in study and control group.
Arm/Group | Multiport Antegrade Cardioplegia | Aortic Root Antegrade Cardioplegia
Serious Adverse Events (participants affected / at risk) | 0/215 | 0/219
Other Adverse Events (participants affected / at risk) | 0/215 | 0/219

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No